CLINICAL TRIAL: NCT04859569
Title: A Phase III Study Comparing Efficacy and Safety of LY01011 and Xgeva®(Denosumab) in Patients With Bone Metastases From Solid Tumors
Brief Title: Efficacy and Safety of LY01011 and Xgeva® in Patients With Bone Metastases From Solid Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY01011/CT-CHN-303
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Bone Metastases From Solid Tumors
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01011 (Experimental): Subcutaneous injection of LY01011 120 mg (1.7ml) every 4 weeks for a maximum of 13 consecutive doses up to week 49.
  Interventions: Drug: LY01011
- Xgeva®+LY01011 (Active Comparator): After subcutaneous injection of Xgeva® 120 mg (1.7ml) every 4 weeks 3 times, patients of Xgeva® group continue to receive LY01011 120 mg (1.7ml) every 4 weeks for ten doses consecutively.
  Interventions: Drug: LY01011; Drug: Xgeva®

INTERVENTIONS:
Drug: LY01011 — subcutaneously (SC) once every 4 weeks (Q4W)
  Other Names: recombinant anti-RANKL human monoclonal antibody injection
Drug: Xgeva® — subcutaneously (SC) once every 4 weeks (Q4W)
  Other Names: Denosumab
  Arms: Xgeva®+LY01011

SUMMARY:
This is a multicenter，randomized, double-blind, active-controlled, parallel-group study comparing efficacy and safety of LY01011 (recombinant anti-RANKL human monoclonal antibody injection) and Xgeva® in patients with bone metastases from solid tumors.

DETAILED DESCRIPTION:
The primary objective is to evaluate the similarity of clinical efficacy between LY01011 and Xgeva® in patients with bone metastases from solid tumors.

The secondary objective is to evaluate the similarity of clinical safety and immunogenicity between LY01011 and Xgeva® in patients with bone metastases from solid tumors.

Each subject will participate in the study for 53 weeks. Treatments are administered on day 1 and Q4W thereafter through week 49. All patients are instructed to take 500 mg calcium and 400 IU vitamin D daily.

ELIGIBILITY:
Inclusion Criteria:

* The subject or his/her guardian and/or impartial witness voluntarily signed the written informed consent form（ICF）.
* Aged 18 to 80 Years old (Female or male subjects to the date of signing the informed consent form).
* Subjects with solid tumor confirmed by histological or cytological examination. At least one documented bone metastasis confirmed by computed tomography[CT], magnetic resonance imaging[MRI]) or pathology (bone biopsy).
* Eastern Cooperative Oncology Group（ECOG）performance status≤2.
* Adequate organ function at baseline.

Exclusion Criteria:

* Prior treatment with denosumab or other RANKL-targeted therapeutic drugs.
* Subjects who previously received any bone-modifying agents (including intravenous or oral bisphosphonates, etc.) for advanced tumor disease.
* Orthopedic surgery or bone-related radiation therapy within 1 month prior to first dose. Bone radioisotope therapy within 6 months prior to first dose, or planned radiation therapy or surgery for bone during the study.
* Past or ongoing osteomyelitis or osteonecrosis of the jaws （ONJ）, an active dental or jaw condition requiring oral surgery, non-healed dental or oral surgery, or any planned invasive dental procedure during the study period.
* Primary central nervous system malignancy. Subjects with central nervous system metastases who have failed local therapy. Subjects with asymptomatic brain metastases or clinically stable brain metastases who do not require steroids and other therapy for brain metastases for ≥ 28 days may be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Natural logarithm change from baseline to week 13 in uNTx/uCr | from baseline to week 13
  Compare LY01011 and Xgeva® for natural logarithm change in bone turnover marker(BTM) -urinary type I collagen cross-linked N-telopeptides (uNTx) corrected for urine creatinine(uCr) in chinese subjects with bone metastases from solid tumors.

SECONDARY OUTCOMES:
The time to first on-study skeletal-related event(SRE) | from baseline to week 53
Incidence of SRE | from baseline to week 53
Percent change in bone specific alkaline phosphatase (s-BALP) from baseline to weeks 13, 25, and 53. | from baseline to weeks 13, 25, and 53
Natural logarithm change in bone turnover marker-uNTx/uCr from baseline to weeks 25 and 53. | from baseline to weeks 25 and 53

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No